## **Coherence Imaging of the Cervical Epithelium**

NCT02903394

Document Date: 17 March 2017

## **Coherence Imaging of the Cervical Epithelium**

Duke PI: Adam WaxDUHS IRB# Pro00070555Jacobi site PI: Michael ZinamanEinstein IRB#: 2016-6643

## Purpose of the Study

The purpose of this study is to develop a multiplexed low coherence interferometry (mLCI) endoscopic probe for mapping the epithelial types of the cervix. This vaginal mLCI probe will obtain optical measurements from the cervix. These measurements can be used to create a map of the surface cells that distinguishes ectocervical epithelia, endocervical epithelia, and the squamocolumnar junction (t-zone) between them, which is the region where cervical dysplasia is most likely to occur.

The research study described here will be a preliminary study to evaluate the performance of the mLCI device for detection of cervical dysplasia. The results from a small study at Duke will help to optimize the function of the mLCI instrument before completing a larger study with collaborators at Jacobi Medical Center (see *Background & Significance* below). The device will be studied in a larger subject population at Jacobi to determine how effectively it can distinguish the types of cervical epithelia.

## Background & Significance

Clinical problem: Cervical cancer, caused by persistent human papillomavirus (HPV) infection, is the second most common female malignancy worldwide. An estimated 500,000 new cases are diagnosed annually, including 12,170 new cases in the U.S in 2012, which reflects an age-adjusted incidence of 8.1 per 100,000 women [1]. Given that cervical cancer typically develops over many years, the early detection of cervical dysplasia (pre-cancers) affords a critical opportunity for treatment and thus prevention of life threatening invasive cancer. In developed countries, the availability of cervical cytology (Papanicolaou smear) for routine screening and colposcopy-directed biopsy for diagnosis has led to decreases in incidence and mortality rates [2]. However, despite their important impact, cytology and colposcopy remain very limited in their sensitivity, specificity, and interobserver reproducibility [3, 4]. The accurate identification of dysplastic areas of the epithelium is challenging and hence clinical guidelines recommend frequent patient screening schedules [5, 6] that are particularly difficult to implement in developing countries. The need for more effective evaluation tools persists.

**Potential Solution:** We propose to address this need by creating an imaging platform that uses *coherence imaging* to evaluate cervical tissues at two length scales. At the millimeter (tissue) scale, a multiplexed LCI (**mLCI**) approach will use multiple imaging channels to efficiently map the cervical epithelium to identify histological structures and red-flag suspicious regions, likely to harbor dysplasia. We have shown that mLCI can survey large areas of tissues *in the female reproductive tract* to obtain diagnostic information on coating by drug delivery gels [7, 8]. Once mLCI identifies suspicious areas, angle-resolved LCI (**a/LCI**) will obtain high resolution, depth resolved nuclear morphology measurements on the micron (subcellular) scale [9, 10]. We have shown that a/LCI can detect dysplastic lesions *in vivo* in the esophagus [11] and *ex vivo* in other types of epithelia such as colon [12] and trachea [13]. The combination of these two optical technologies, mLCI and a/LCI, will provide a unique platform for comprehensive assessment of the cervix at both tissue and subcellular scales. The novel technology will impact clinical detection of cervical dysplasia as well as support clinical and translational research on the fundamental biology of the cervical epithelium.

Rationale for collaborative project: The Duke team has had significant success in developing endoscopic imaging modalities for detection of precancerous tissues. Ongoing collaboration between the group in Duke BME and the Department of Ob/Gyn at Duke University Medical Center (DUMC) has produced important studies of the pharmacology of anti-HIV microbicides delivered to the lower female reproductive tract [7, 8, 14-17]. Here we seek to forge a broader collaboration to bring together the established team at Duke with a leading group in clinical research at Jacobi Medical Center. Jacobi serves a predominately minority population, and due to the largely immigrant status of women over age 26, HPV vaccination rates are low. Therefore, it has a large population of women with HPV-associated cervical dysplasia and a significant number of women with cervical cancer.

This collaboration will create a powerful combination of technology development and translation at the leading edge of gynecological biomedicine. This project will develop and test new instruments for cervical imaging at Duke and field test these technologies in the large, diverse patient population available at Jacobi Medical Center. The anticipated outcome is the creation of a diagnostic imaging tool that can screen women for cervical precancers and cancers and/or triage precancerous lesions in women who have had a positive cytology test.

#### **INNOVATION**

Novel multimodal imaging platform that combines mLCI and a/LCI: The mLCI technology is unique in its ability for depth resolved imaging of wide areas of tissues. While LCI can obtain high resolution tomographic images at micron scales, as is done in optical coherence tomography (OCT), that approach is limited by often cumbersome scanning mechanisms and the large volume of data generated. Instead, mLCI uses sparse sampling and multiple parallel channels to more efficiently scan wider tissue areas. We will exploit this ability to create a new modality for quickly mapping the cervical epithelium, analogous to the function of colposcopy, but with improved performance. This is a particular challenge due to the complex combination of cervical epithelial types that are often in transitional states (columnar to metaplastic to squamous). As a counterpart to the mLCI, the a/LCI modality will combine the depth resolution and penetration of OCT with the sensitivity to subcellular structure that is obtained via light scattering, providing a function analogous to biopsy. Our group has recently validated a/LCl as an in vivo method for identifying dysplastic esophageal tissues [11]. Although prior research has applied OCT and light scattering to cervical dysplasia [18, 19] these approaches have not been clinically feasible. The unique capabilities of a/LCI, which enable high accuracy in detecting dysplasia, offer a significant potential for clinical translation. By combining mLCl and a/LCl into a single integrated platform, we will capitalize on recent trends in multimodal imaging. As identified by clinicians and researchers in multiple fields [20, 21], optimal screening methods can be realized by using a wide area scan to survey for suspicious regions in tandem with a high resolution modality to further diagnose those regions. Thus, we will implement this paradigm and create a hybrid imaging modality that integrates tissue and cellular imaging data. The unique power of this multimodal LCI device will lie in its ability to accurately identify dysplastic and cancerous tissues against the background of the complex tissue types that comprise the cervical epithelium.

Innovation in clinical care of cervical disease: In the clinic, the clear advantage of the multimodal LCI platform will be its ability to support clinical decision-making without relying on gross clinical colposcopic impression, the traditional but somewhat subjective diagnostic method. Further, the potential to provide reliable "real-time" information to the clinician would allow immediate treatment of epithelial abnormalities. We expect this

device to be uniquely applicable to women of all ages in contrast to the recent implementation of screening biomarkers such as HPV DNA testing which are restricted to older women. Our field trials will access the diverse patient population found at Jacobi OB/GYN. This population represents the full spectrum of cervical health, including healthy young women and those with incident HPV infection, persistent HPV infection, benign cervical lesions, cervical precancers, and cancer. Our proposal to develop an accurate and efficient tool for cervical cancer screening will rely on its ability to detect disease in the setting of complex tissue compositions inherent to the cervix—the downfall of many prior optical technology attempts. Innovation is inherently risky; however our combined expertise in coherence imaging and the clinical study of the cervical epithelium will support the success of the proposal.

### Multi-site Study: Responsibilities

Dr. Wax, the Duke PI of this study, is the primary awardee of the NIH grant supporting this work. Dr. Wax and his team have developed the mLCI research device and will conduct a small study at Duke (described below) to assess if any adjustments to the device are needed before it is sent to Jacobi Medical Center for the larger study. The study at Jacobi Medical Center will be funded as a subaward / consortium agreement of Dr. Wax's NIH grant. The research proposed in this study protocol addresses Specific Aim 1 of the NIH grant.

Duke will recruit up to 15 women to enroll in this study, in order to achieve the target number of 10 subjects who complete the study at that site. Jacobi will enroll up to 100 women for this study, in order to achieve the target number of 40 women who complete the study at that site. Data from both sites will be analyzed at Duke. Data received from Jacobi will be de-identified before being sent to Duke. Study conduct at Duke will be under the oversight of the IRB of the Duke University Health System. Study conduct at Jacobi Medical Center will be under the oversight of the IRB of the Albert Einstein College of Medicine and Montefiore Medical Center.

#### **Design & Procedures**

#### **mLCI** instrument

The purpose of this instrument is to obtain optical measurements from the cervix via a vaginal probe to create a map of the surface cells that distinguishes the ectocervical and endocervical epithelia. The boundary between the two cell types is known as the squamocolumnar junction, or "t-zone", which is the transitional region at which cervical dysplasia is most likely to occur.

The instrument delivers infrared light to 36 locations on the cervix, and measures the depth-profile of back-scattered light from each location using low coherence interferometry (LCI). This technique is thus termed multiplexed LCI (mLCI). The LCI profile data is stored by a computer for subsequent analysis to identify cell type.

The components of the mLCI instrument are grouped in the following modules: 1) Optical probe, 2) mLCI interferometer, 3) white light imaging module, 4) computer, and 5) physical enclosure.

#### **Optical Probe**

The optical probe is primarily cylindrical in form, with a diameter of approximately 25 mm and a rigid length of approximately 270 mm. The probe housing is fabricated by a 3D printing process known as fused deposition modeling (FDM). The material is MED-610 (Stratasys Inc., Eden Prairie, MN), a transparent polymer certified as biocompatible.

The adhesives used on the external seams of the probe are Silastic Medical Adhesive Type A (Dow Corning, Midland, MI), a soft silicone adhesive. A 36-channel single-mode fiber bundle is contained within the probe housing, as well as several glass optical elements for imaging. The rounded tip of the probe is intended to contact the cervical surface, and the focus of mLCI imaging is located on the plane of this tip.

The probe also contains fiber optics that deliver white LED illumination to the region of imaging and collects wide-field imaging information through a fiber bundle to provide real-time video endoscopic guidance for probe placement.

A flexible tether containing the 36-fiber bundle and white light optical fibers protrudes from the proximal end of the probe and is connected to the mLCI interferometer and white light imaging modules, respectively.

The full length of the probe is not intended for vaginal insertion. A demarcation line approximately 220 mm from the probe tip indicates the line beyond which the probe should not be inserted. High-level disinfection procedures as described in this document will be performed up to the line.

The probe contains no electrical components or wires.

#### mLCI interferometer

The centerpiece of LCI instrumentation is an interferometer, in which light from a known reference distance is combined with light returning from the probe. In our multiplexed design, 6 channels are simultaneously illuminated and interfered with each of 6 independent references. The mLCI thus contains 6 complete fiber optic interferometers, and fiber-optic switches redirect the optical inputs and outputs to progress through the 36 channels in a sequence of 6 acquisitions.

The 6 interferometers in the mLCl system are connected individually to each of 6 parallel fiber-optic spectrometers (Avantes, Broomfield, CO), which interface with the computer via one common USB connection.

The light source from the mLCI system is a superluminescent diode (Superlum, Moscow, Russia) emitting infrared light at wavelengths between 815 and 845 nm. The total output power of the SLD at its output aperture is less than 25 mW, but the amount of power delivered by the probe is far less. The power at each of the individual 36 foci at the probe output is less than 500  $\mu$ W (0.5 mW).

The maximum permissible exposure (MPE) for exposures greater than 10 seconds on skin is 3.6 mW/mm² at our principal wavelength of 830 nm (ANSI Z136.1). In our system, only 6 channels are simultaneously illuminated. Our imaging region in the tissue is 16 mm (defined by the length of our row of 6 spots)  $\times$  3.5 mm (defined by the minimum limiting aperture given in ANSI Z136.1) = 56 mm². Our total permissible power is thus 3.6 mW/mm² x 56 mm² = 201 mW. The totality of our 6 foci = 6 x 0.5 mW = 3 mW, which is far short of the ANSI MPE.

#### White light imaging module

A white light imaging module is configured to provide video endoscopy guidance for the probe placement on the cervix. This module consists of a white light LED optically coupled to an illumination fiber that is enclosed in the probe, as well as an imaging

camera and relay optics to digitize the endoscopic image from the probe's white light fiber bundle.

#### Computer

A laptop computer (Lenovo, Beijing, China) performs the data acquisition and control through a custom application in Labview (National Instruments, Austin, TX). Real-time display of the white-light endoscopic images is provided, as well as synchronized acquisition of LCI data from spectrometers. Through a customized microcontroller module, this software also implements control of reference mirror positions by stepper motor and control of fiber-optic switch positions.

## Physical enclosure

The mLCI interferometer, white light imaging module, and computer are situated upon a wheeled steel cart. The fiber-optic interferometer components are protected by a metal enclosure. Power to all components is provided through standard 120V mains routed through an uninterruptible power supply (UPS), which allows temporary disconnection of AC power for system transportation or due to accidental action without interrupting the operating state of the mLCI system.

### Study Procedures for subjects at Duke

Each subject will attend 1 study visit that will last between 1 - 1.5 hours and include the following procedures.

- Read consent form
- Ask / answer questions
- Sign consent form
- Complete brief medical questionnaire to determine eligibility
- Urine pregnancy test must be negative before imaging can occur
- mLCl examination of the cervix (without speculum)
- mLCl examination of the cervix (with speculum)

We will obtain written informed consent and confirm eligibility criteria. Data collection will include a brief medical history and pregnancy testing. Participants will be interviewed one-on-one to complete the questionnaire regarding medical and reproductive history. The nurse or doctor will then perform the mLCI study measurements.

The nurse or doctor will gently place the mLCI probe against the cervix. Lubricant will be placed on the outside of the probe for subject comfort. White light camera visualization, incorporated into the mLCI probe, will guide the probe positioning by the clinician to confirm contact with the cervical epithelium. Up to 4 minutes will be allotted for probe manipulation for optimal contact. The probe will then be held in place for mLCI data acquisition for up to 1 minute. When data collection is completed, or permitted time is elapsed, the mLCI probe will be removed and placed on a custom holder that prevents the contact portions of the probe from coming into contact with contaminating surfaces.

The nurse or doctor will then insert a speculum in order to directly visualize the cervix. The mLCI probe will again be placed against the cervix with 4 minutes allotted for probe manipulation and 1 minute for mLCI measurements.

If manipulation of the probe with the aid of a speculum does not allow satisfactory placement on the cervix for mLCI imaging within the permitted time, an additional attempt may be made with an alternate speculum, such as a Pedersen Open-Sided speculum, if

the medical practitioner performing the procedure believes the alternate speculum to be more likely to result in correct probe placement. If the alternate speculum is used, then an additional 4 minutes will be allotted for probe manipulation with the alternate speculum, and 1 minute for mLCI measurements. The timing of each phase of the procedure is summarized in the following table.

**Table 1**: Maximum allotted times of mLCl probe insertion

| Insertion<br>method | Criteria | Time for probe placement | Time for mLCl acquisition | Maximum total time |
|---|---|---|---|---|
| Without speculum | All patients | 4 min | 1 min | 5 min |
| With standard speculum | All patients | 4 min | 1 min | 5 min |
| With alternate speculum | Optional (only if standard speculum not satisfactory AND practitioner believes alternate may achieve better result) | 4 min | 1 min | 5 min |

Comparing measurements made by inserting the mLCI device with and without a speculum will allow us to determine if the white light visualization by the camera is sufficient to correctly place the probe over the cervix without having to use a speculum in future studies. The ability to use an alternate in the event that a conventional speculum does not permit adequate mLCI probe placement will also inform our selection of the type of speculum, if any, that is most suited for subsequent studies.

### Study Procedures for subjects at Jacobi

Subjects will be informed of the study when they present to the clinic for a regular clinical care visit. If interested in participating, subjects will complete the following study-related procedures in addition to the standard of care visit procedures.

- Read consent form
- Ask / answer questions
- Sign consent form
- Urine pregnancy test must be negative before imaging can occur
- Colpophotography of cervix to compare with mLCI data
- mLCl examination of the cervix (with speculum)

We will obtain written informed consent and confirm eligibility criteria. Data collection will include a brief medical history and pregnancy testing.

The doctor will then insert a speculum in order to directly visualize the cervix. Colpophotographs will be taken to compare to mLCl data during data analysis. The doctor will then gently place the mLCl probe against the cervix. White light camera visualization, incorporated into the mLCl probe, will guide the probe positioning by the clinician to confirm contact with the cervical epithelium. The probe will then be held in place for mLCl data acquisition for up to 1 minute. When data collection is completed, the mLCl probe will be removed and placed on a custom holder that prevents the contact portions of the probe from coming into contact with contaminating surfaces.

The doctor will then continue with the rest of the patient's standard of care visit procedures.

At some visits, the physician may choose to make an additional measurement with the mLCI device, by inserting it without a speculum and using the white light camera (incorporated into the mLCI probe) for visual guidance to position the probe. Comparing measurements made by inserting the mLCI device with and without a speculum will allow us to determine if the white light visualization by the camera is sufficient to correctly place the probe over the cervix without having to use a speculum in future studies.

#### **Selection of Subjects at Duke**

This project will recruit healthy women who:

- are able to provide informed consent
- are at least 21 years old
- are willing to abstain from sexual intercourse for at least 24 hours before the study visit

Participants meeting any of the following exclusion criteria will be excluded from taking part in this study. Women must not:

- be pregnant
- have given birth to a baby
- have a current gynecologic infection or discharge
- be using an IUD
- have had any cervical surgery
- have had medical or cosmetic surgery involving the reproductive organs or genitals within the past 6 months
- be currently enrolled in any research studies involving the application of vaginal formulations
- be employed or supervised by the study investigators
- have any other condition that, in the opinion of the study clinician, would contraindicate participation in the study

#### **Selection of Subjects at Jacobi**

We do not have any role in selection of the research subjects at Jacobi: this is the responsibility of that site.

#### **Subject Recruitment & Compensation at Duke**

We will recruit up to 15 women to enroll in this study, in order to achieve the target number of 10 subjects who complete the study.

The study will be advertised on the ResearchMatch website. Recruiting will be managed by our study coordinator. The inclusion of minorities in the group of women recruited will reflect the local distribution in the Durham area.

After learning about the study, prospective subjects will call the study coordinator for more information. During this telephone call, the study coordinator will state the study requirements plus a brief description of the procedures. If the prospective subject is interested in participating in the study, a study visit will be scheduled. The prospective subject's contact information will be kept in a locked desk or file cabinet or password protected file in the study coordinator's office. If the prospective subject states that she does not qualify or is not interested in participating, the contact information will be destroyed.

Subjects will be compensated \$50 per visit (1 visit per subject).

### **Subject Recruitment & Compensation at Jacobi**

We do not have any role in recruiting or compensating research subjects at Jacobi: this is the responsibility of that site.

## **Consent Process at Duke**

The consent process will be conducted by the study coordinator at a meeting in the study coordinator's office or other suitable private location (PI's office, conference room, clinic consult room).

Thirty minutes will be allocated for conducting the initial consent discussion, allowing time for the prospective subject to read the consent form and ask any questions she may have. At the consenting interview, the study coordinator will:

- explain the study procedures in detail, including risks and compensation
- inform the participant of her rights as a research subject, including the right to withdraw at any time
- give the participant a chance to ask any questions she may have

The prospective subject may then sign and date the consent form if she chooses to participate at that time. She may take more time to consider her decision and sign the consent form at a later date if she chooses. The prospective subject will have as much time as she needs to decide whether or not to participate. However, enrollment will continue, and if all study slots are full by the time the prospective subject decides to participate, she may not be enrolled in the study. Once the consent form is read and signed, the subject and study coordinator will complete the Informed Consent Review Check Sheet to document the consent process.

The prospective subject will then complete a brief screening questionnaire and a urine pregnancy test. Results from the screening questionnaire and pregnancy test will be reviewed to determine if the subject is eligible to continue participation in the study. If the screening test indicates pregnancy, the participant will be excused from the study and advised to follow up with her physician. Subjects who pass screening will be enrolled in the study on a first-come, first-served basis.

The prospective subject may ask questions at any time by calling the study coordinator or PI. The study coordinator will conduct all consent discussions and study visits and will be available to answer any questions that arise at those times.

To minimize the possibility of coercion or undue influence, study personnel will inform subjects of their rights as a research participant, including their right to refuse to participate or to withdraw from the study at any time without penalty. Reimbursement (\$50 per session) is not believed to be coercive, based on the time required and the nature of the research. The amount of reimbursement is comparable to similar studies. Duke students and employees under direct supervision of the study staff will not be allowed to participate in this study.

Since recruiting materials (website postings) are in written English, it is expected that anyone who calls to inquire about participating in the study will be able to read English. No provisions are in place for potential participants who do not understand English.

#### **Consent Process at Jacobi**

We do not have any role in consenting subjects at Jacobi: this is the responsibility of that site.

## Subject's Capacity to Give Legally Effective Consent at Duke

Subjects who do not have the capacity to give legally effective consent will not be included in this study.

## Subject's Capacity to Give Legally Effective Consent at Jacobi

We do not have any role in assessing subjects' capacity to give legally informed consent at Jacobi: this is the responsibility of that site.

#### **Study Interventions**

See above.

## Risk/Benefit Assessment of the study in general

#### Potential Risks

Potential risks include:

- 1. breach of confidentiality
- 2. coercion
- 3. discomfort with the nature of the research
- 4. side effect from study procedures and/or devices

#### Potential Benefits

There is no direct benefit to subjects participating in this research study. However, the novel mLCI device to be developed in this proposal would potentially advance the management of cervical dysplasia by assisting clinical decision-making without relying on gross colposcopic impression. The current proposal is to conduct the early feasibility studies necessary for technology development. Data will also be collected about epithelial characteristics as visualized by mLCI, which could improve our understanding about the basic biology of the cervical epithelium. The long-term goal is to develop devices that could be incorporated into routine clinical care. The mLCI device could provide real-time information to the clinician and reduce the number of clinical visits needed.

#### Alternative Treatments

There are no alternative treatments to participating in this research. It is not intended to be therapeutic, but to acquire basic scientific knowledge.

# Risk Assessment and Risk Minimization for Study Activities at Duke Potential Risks

Potential risks include:

- (1) breach of confidentiality
- (2) coercion
- (3) discomfort with the nature of the research
- (4) side effects from study procedures and/or devices

## **Breach of Confidentiality**

Subjects will provide personal information, including sexual history and health information. Breach of confidentiality will be avoided by training research staff in the protection of human subjects and by coding and limiting access to data. Each participant will be assigned a research subject number. The only documents linking the

subject's identity with her subject number will be the consent form and the enrollment log. The contact information list and payment request forms will contain the subject's identity only. The medical questionnaire, pregnancy test result, and data spreadsheets will reference the subject number only. The subject's social security number, required on the payment request form, will be blacked out once payment has been processed. Once the study is complete, all contact information will be deleted, unless the participant requests to be contacted for future studies conducted by Dr. Wax or his colleagues. All of the participant's study documents will be kept in a locked file cabinet in the study coordinator's office. Databases containing PHI will be maintained on a password-protected computer with full disk encryption.

#### Coercion

Coercion occurs when potential participants feel compelled to participate in research for reasons such as perceived demand or the availability of large sums of reimbursement. This can be particularly true when there is little benefit to the individual for their participation. In this study, there is minimal risk of coercion as personnel will inform subjects of their rights as a research participant, including their right to refuse to participate or to withdraw from the study at any time without penalty. Reimbursement (\$50) is not believed to be coercive, based on the time required and the nature of the research. The amount of reimbursement is comparable to similar studies.

#### Discomfort with the Nature of the Research

Participants may feel discomfort with the personal nature of this research. Before the participant is enrolled in the study, detailed study procedures will be explained so she is aware of what the research entails. Subjects will provide personal information, such as sexual health and history. Some study procedures will be conducted with the physician/nurse and research assistant/chaperone in the room, including insertion of the mLCI device into the vagina by the physician/nurse (similar to a pelvic exam) and making measurements with the device. Participating in these research procedures and providing personal information may be uncomfortable for some women. It is unlikely this discomfort will result in any serious adverse events. Should participants report discomfort with the research, they will be reminded of their rights to not participate in the study or to withdraw from the study at any time. Subjects may contact the principal investigator or one of the study physicians at any time to discuss questions or concerns about the study.

## Side Effects from Study Procedures and/or Devices

Risks of the mLCI Device: The mLCI device will be handled gently for placement against cervical tissue. We expect very minimal risk for tissue abrasion or irritation as the devices will have a smooth plastic and silicone surface and commercial gynecological lubricant will be applied before cervical contact. The device will be cleaned in full accordance with high level disinfection clinical procedures at DUHS. Specifically, probes will be enclosed in a Trophon EPR high-level disinfection system to disinfect all external surfaces. Study staff will complete training and competency reviews per institutional procedures. For the mLCI technique, a fiber optic bundle transmits near infrared light onto the epithelia to image the cervix. The light source has been either certified for medical use or tested to demonstrate that it complies with medical safety standards.

## Costs to the Subject at Duke

There will be no costs to the subject as a result of participating in this study.

## **Data Analysis & Statistical Considerations**

## Data analysis for Duke site

The proposed study is designed as a pilot study, intended to provide feasibility and usability data to inform future studies on a larger scale. The planned pilot study will include 10 subjects, which will yield success/failure metrics of the probe design with 10% precision. Elements of the probe performance that will be evaluated include ease of use by the medical practitioner, patient comfort, ability to access the relevant anatomy, and quality of mLCI imaging data. Because the goal of the pilot study is the evaluation of general feasibility, no subject data will be excluded if no predetermined exclusion criteria are met.

#### Data analysis for Jacobi site

Construction of epithelium maps by mLCI: Maps of the cervix delineating the T-zone will be created from each subject's mLCI data. The extent of columnar and squamous epithelia will be reported as a percentage of the image of the epithelium. Each scan in the 36 point field will initially be reviewed manually to determine the epithelium type based on the depth-resolved reflection profile for that point. The presence of clear histological layers in indicative of squamous epithelium while a thinner layer with less structure indicates columnar epithelium [22]. As we compile a database of mLCI maps of the cervix, we will develop automated algorithms for assessing epithelial types and transitions by using cluster analysis to discriminate scans. The mLCI maps will be compared to digital colpophotography analysis to assess accuracy.

Measurement of epithelial areas by colpophotography: Digital colpophotographs will be viewed in Adobe Photoshop for quantitative computerized planimetry as previously published [23, 24]. We will manually outline all areas of columnar, metaplastic and squamous epithelia and the total visible cervical face. Total pixel counts of the various epithelial types will be calculated and ectopy expressed as percentage of the total cervix.

Correlation of mLCI images to colpophotographs and detailed written maps: The mLCI epithelial maps will be visually compared to colpophotographs to achieve co-registration. This is feasible based on the relatively modest number of patients in the study. The written map and white light imaging via the probe will aid in coregistration. We will correlate mLCI readings with calculated areas of epithelial types (pixel counts and percentage). Biostatistical analyses will address covariates including age, infections, cytology, menstrual cycle, and sexual behaviors.

Potential problems, alternative strategies, and benchmarks for success: The mLCl approach will be viewed as successful if there is less than average absolute difference of 10% in the area estimate compared with manual analysis.

#### **Data & Safety Monitoring**

#### Reporting of Adverse Events

An adverse event is defined as any untoward medical occurrence in a clinical research subject participating in the clinical study of the mLCI device. Any AE that occurs between the time a study participant signs the informed consent form and the time she departs the study at the end of the imaging session will be captured and recorded. Study participants will be instructed to contact the study site staff to report any AEs they may experience after completion of their participation. AE resolution will consist of evaluating instrument design and application to assess the potential source and implementing design changes

to mitigate the risk of further AE. If necessary, AEs will be reported to the IRB according to IRB guidelines.

## Safety Monitoring

During the proposed trial of the mLCI device, weekly status reports will be submitted to the Duke PI from the Jacobi site. These reports will include all adverse events reported for the study, determined to be related or unrelated to the study protocol. The study team will meet, as needed, throughout the period of study to review any reported adverse events and address any potential safety concerns.

## Data accuracy and protocol compliance

Data acquired during the clinical study will be reviewed on a weekly basis by Duke lab personnel to assess if the data appear to be consistent with expected operating characteristics of the device. In the event that data do not appear satisfactory, a review of protocol compliance will be conducted. If the protocol has been followed, a technical inspection of the device by Duke lab personnel will be scheduled and further study will be suspended until instrument function has been verified.

## Privacy, Data Storage & Confidentiality at Duke

The investigator will ensure that the subject's anonymity is maintained. Subjects will not be identified in any publicly released reports of this study. All records will be kept confidential to the extent provided by federal, state and local law. The study monitors and other authorized representatives of the Sponsor may inspect all documents and records required to be maintained by the Investigator, including but not limited to, medical records. The investigator will inform the subjects that the above-named representatives will review their study-related records without violating the confidentiality of the subjects. All laboratory results, evaluation forms, reports, and other records that leave the site will be identified only by a coded number in order to maintain subject confidentiality. Clinical information will not be released without written permission of the subject, except as necessary for monitoring by the IRB, the FDA, the NIH, the OHRP, or the sponsor's designee.

Due to the personal nature of this research, all subject interviews will take place in a private office and all study visits will take place in a private clinic room. Some study procedures will be conducted with the physician/nurse and research assistant/chaperone in the room, including insertion of the LCI device into the vagina by the physician/nurse (similar to a pelvic exam) and making measurements with the device. The subject will be draped with a sheet during these study procedures to provide as much privacy as possible.

Subjects will provide personal information, including sexual history and health information. All study personnel will complete training in the conduct of human subjects research in order to protect against possible breach of confidentiality. Identifiers will be removed from any data being analyzed. Each participant will be assigned a research subject number. The only documents linking the subject's identity with her subject number will be the consent form and the enrollment log. The contact information list and payment request forms will contain the subject's identity only. The medical questionnaire, pregnancy test result, and data spreadsheets will reference the subject number only. The subject's social security number, required on the payment request form, will be blacked out once payment has been processed. Once the study is complete, all contact information will be deleted or destroyed, unless the participant requests to be contacted for future studies conducted by Dr. Wax or his colleagues.

All of the paper study documents will be kept in a locked file cabinet in the study coordinator's office. Electronic study records will be maintained on a password-protected computer with whole disk encryption in the study coordinator's office. To protect against the possibility of loss of research records, database files will be periodically backed up to a DUHS network drive.

#### References

- 1. Howlader, N., et al. SEER Cancer Statistics Review, 1975 2009 (Vintage 2009 Populations). 2012 April; Available from: http://seer.cancer.gov/csr/1975 2009 pops09/.
- 2. Gustafsson, L., et al., *International incidence rates of invasive cervical cancer after introduction of cytological screening.* Cancer Causes Control, 1997. **8**(5): p. 755-63.
- 3. Chase, D.M., M. Kalouyan, and P.J. DiSaia, *Colposcopy to evaluate abnormal cervical cytology in 2008*. Am J Obstet Gynecol, 2009. **200**(5): p. 472-80.
- 4. Stoler, M.H. and M. Schiffman, *Interobserver reproducibility of cervical cytologic and histologic interpretations: realistic estimates from the ASCUS-LSIL Triage Study.* JAMA, 2001. **285**(11): p. 1500-5.
- 5. ACOG Practice Bulletin no. 109: Cervical cytology screening. Obstet Gynecol, 2009. 114(6): p. 1409-20.
- 6. Wright, T.C., Jr., et al., 2006 consensus guidelines for the management of women with abnormal cervical cancer screening tests. Am J Obstet Gynecol, 2007. 197(4): p. 346-55.
- 7. Drake, T.K., et al., Design and validation of a multiplexed low coherence interferometry instrument for in vivo clinical measurement of microbicide gel thickness distribution. Biomedical Optics Express, 2011. **2**(10): p. 2850-2858.
- 8. Drake, T.K., et al., *In vivo optical imaging of human vaginal gel thickness distributions with a probe-based, dual-modality instrument.* J Biomed Opt, 2012. **17**(11): p. 116014.
- 9. Chalut, K.J., W.J. Brown, and A. Wax, *Quantitative phase microscopy with asynchronous digital holography*. Opt Express, 2007. **15**(6): p. 3047-52.
- 10. Wax, A., et al., Cellular organization and substructure measured using angle-resolved low-coherence interferometry. Biophys J, 2002. **82**(4): p. 2256-64.
- 11. Terry, N.G., et al., *Detection of dysplasia in Barrett's esophagus with in vivo depth-resolved nuclear morphology measurements.* Gastroenterology, 2011. **140**(1): p. 42-50.
- 12. Terry, N., et al., *Detection of intestinal dysplasia using angle-resolved low coherence interferometry*. J Biomed Opt, 2011. **16**(10): p. 106002.
- 13. Chalut, K.J., et al., *In situ assessment of intraepithelial neoplasia in hamster trachea epithelium using angle-resolved low-coherence interferometry*. Cancer Epidemiol Biomarkers Prev, 2007. **16**(2): p. 223-7.
- 14. Geonnotti, A.R. and D.F. Katz, *Dynamics of HIV neutralization by a microbicide formulation layer: Biophysical fundamentals and transport theory.* Biophysical Journal, 2006. **91**(6): p. 2121-2130.
- 15. Henderson, M.H., et al., *Optical imaging and analysis of human vaginal coating by drug delivery gels.* Contraception, 2007. **75**(2): p. 142-151.
- 16. Lai, B.E., et al., Transport Theory for HIV Diffusion through In Vivo Distributions of Topical Microbicide Gels. Biophysical Journal, 2009. 97(9): p. 2379-2387.
- Lai, B.E., et al., Dilution of microbicide gels with vaginal fluid and semen simulants: Effect on rheological properties and coating flow. Journal of Pharmaceutical Sciences, 2008. 97(2): p. 1030-1038
- 18. Georgakoudi, I., et al., *Trimodal spectroscopy for the detection and characterization of cervical precancers in vivo*. Am J Obstet Gynecol, 2002. **186**(3): p. 374-82.
- 19. Mourant, J.R., et al., *In vivo light scattering measurements for detection of precancerous conditions of the cervix.* Gynecol Oncol, 2007. **105**(2): p. 439-45.
- 20. Peery, A.F. and N.J. Shaheen, *Optical coherence tomography in Barrett's esophagus: the road to clinical utility.* Gastrointest Endosc, 2010. **71**(2): p. 231-4.
- 21. Thekkek, N. and R. Richards-Kortum, *Optical imaging for cervical cancer detection: solutions for a continuing global problem.* Nat Rev Cancer, 2008. **8**(9): p. 725-31.

- 22. George, M., et al., Optical coherence microscopy for columnar and squamous epithelium discrimination: Potential and clinical applicability, in Cars 2001: Computer Assisted Radiology and Surgery, H.U. Lemke, et al., Editors. 2001, Elsevier Science Bv: Amsterdam. p. 1023-1028.
- 23. Hwang, L.Y., et al., Factors that influence the rate of epithelial maturation in the cervix in healthy young women. J Adolesc Health, 2009. **44**(2): p. 103-10.
- 24. Moscicki, A.B., et al., *The significance of squamous metaplasia in the development of low grade squamous intraepithelial lesions in young women.* Cancer, 1999. **85**(5): p. 1139-44.